CLINICAL TRIAL: NCT04124835
Title: Effectiveness of Using the Swiss Ball in Birth Compared to Habitual Care on Maternal and Neonatal Outcomes: Randomized and Pragmatic Clinical Trial
Brief Title: Effectiveness of Using the Swiss Ball in Birth
Acronym: BIRTHBALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Principal Investigator, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BIRTHBALL
Record Dates: First submitted 2019-10-03; First posted 2019-10-11 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Labor Pain
Keywords: Labor, Obstetric; Physical Therapy Modalities
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: This will be a randomized, open-label study aimed at evaluating the effectiveness of using the Swiss Ball, without comparing it with usual care in maternal and neonatal outcomes. Patients will be randomized to receive standard care, as the ward is already a humanized, position-free approach, and to press or join all of this standard product, receive guidance on the use of the Swiss Ball.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, the use of the Swiss Ball will be performed through active exercises of pelvic anteversion and retroversion, lateralization and circumduction according to the obstetric evaluation.
  Interventions: Other: Swiss Ball
- Control Group (Other): The control group will receive the usual routine care of the service.
  Interventions: Other: Control Grup

INTERVENTIONS:
Other: Swiss Ball — Top narrow (DeLee Plan -5 to -1 or Hodge Plan 1-3) Retroversion, lateralization and pelvic circumference exercises with abducted hips and external rotation will be encouraged. Exercises according to fetal positioning: Four ball-assisted supports and / or biped stance with anterior trunk inclination with asymmetrical opening of lower limbs with the aid of the ball. The hips will be in abduction and external rotation.
  Lower Narrow (DeLee Plan +1 to +5 or Hodge Plan 3-4) Pelvic anteversion, tilt, and circumference exercises with abducted hips and internal rotation will be encouraged. Exercises according to fetal positioning: Four ball-assisted supports and / or biped stance with anterior trunk inclination with asymmetrical opening of lower limbs with the aid of the ball. The hips will be in abduction and internal rotation.
  Arms: Intervention Group
Other: Control Grup — Habitual Care of the Service.
  Arms: Control Group

SUMMARY:
A randomized clinical trial will be conducted to evaluate the effectiveness of using the Swiss Ball as a resource that reduces the length of labor time. The study will be conducted in the Low Risk Labor and Delivery sector of (Instituto Materno Infantil Professor Fernando Figueira) IMIP, which has a team of obstetric nurses, medical coordination and physical therapy support. The study population will be composed of low risk parturients admitted to the sector. Parturients who meet the inclusion criteria after signing the Informed Consent Form will be allocated into two groups: Group A (experimental) and Group B (control). Group A will be encouraged to use the Swiss Ball through pelvic movements, and Group B will go through the usual routine. Study results will be evaluated by assistants during labor and immediately after delivery.

DETAILED DESCRIPTION:
Background: The Birth Ball, in childbirth care, has become a widely used resource in obstetrical centers, as it allows the adoption of vertical postures and exercises of pelvic mobility. It is an inexpensive and user-friendly feature that can facilitate pelvic exercise and thus contribute to positive maternal and neonatal outcomes.

Aim: To evaluate the effectiveness of the use of the Birth Ball compared to usual care in reducing the time of the first period of labor.

Methods: This is a randomized and pragmatic clinical trial that will be developed at the IMIP Childbirth Center in the state of Pernambuco. Pregnant women with normal risk, will be included in the first period of labor, with term gestation of the single and cephalic fetus, and pregnant women with a fetus dead, with a psychiatric disorder, using psychoactive drugs and in use of epidural analgesia or oxytocin prior to randomization. The sample size was calculated in 200 parturients, being randomly allocated 100 pregnant women for the experimental group and 100 for the control group, according to a list of random numbers specifically generated for this purpose. The duration of the first period of labor and, as secondary, pain, duration of the second period, birth routes, use of analgesia and oxytocin before randomization, fatigue, anxiety, maternal satisfaction, APGAR in the 5th neonatal resuscitation and hospitalization in a neonatal intensive care unit. The intervention group will use Birth Ball to perform active anteversion and pelvic retroversion exercises, lateralization and circumference according to the obstetric evaluation. The control group will receive the usual routine care of the service. Measurements will be made during and after fetal birth. The control group will receive the usual routine care of the service. Measurements will be made during and after fetal birth. To compare the continuous variables, the mean difference with the 95% Confidence Interval and Student's t-Test will be used. In order to compare the dichotomous variables, the Chi-square Test will be used. The Relative Risk will be calculated with the respective Confidence Interval of 95%. Data analysis will be performed using the Epi Info for Windows, version 3.5.4. The data will be presented in tables.

Ethical aspects: This study will comply with Resolution 466/12 of the National Health Council and will be submitted to the IMIP Research Ethics Committee, beginning only after its approval. All participants will only be included if they voluntarily agree to participate by signing the Free and Informed Consent Form. The research protocol will be registered in Clinical Trials.gov.

There are no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman in the first period of active labor;
* usual risk pregnancy;
* Single fetal pregnancy in cephalic presentation.

Exclusion Criteria:

* Pregnancy with dead fetus;
* Pregnant women with cesarean section indicated upon admission or until the time of approach;
* Pregnant women with limited mobility;
* Pregnant women with hip and pelvic fractures presenting difficulties in sitting position;
* Use of psychoactive drugs;
* Use of epidural analgesia or oxytocin before randomization.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Length of the first period of labor | 12 hours
  Duration in minutes of the first period of labor: that will be considered from the time of admission with active labor (at least 3 contractions every 10 minutes associated with cervical dilatation of at least five centimeters), until complete dilation and urge to push

SECONDARY OUTCOMES:
Length of the second period of labor | 5 hours
  Duration in minutes of the second period: second period will be considered from the that complete dilation and spontaneous pushes start, until delivery of the baby
Maternal pain | 30, 60 and 90 minutes
  The level of pain reported by the patient at each assessment (30, 60 and 90 minutes of use of the Swiss Ball), ranging from zero to ten, with zero being considered the total absence of pain and ten the most extreme, unbearable pain, never before felt. throughout life. Evaluated by visual analog scale (VAS)
Severe Perineal laceration | 1 hour postpartum
  Rate of severe perineal laceration (including third and fourth degree laceration)
Rate of episiotomy | 1 hour postpartum
  Incidence of episiotomy (incision made in the perineum -muscle area between the vagina and anus- to enlarge the birth canal with the theoretical objective of preventing irregular laceration during the passage of the baby. It may be median or mid-lateral.
Type of delivery | 1 hour postpartum
  Frequency of the type of birth, which may be: vaginal, instrumental birth (assisted with forceps or vacuum extraction) or cesarean.
Instrumental birth | 1 hour postpartum
  Incidence of instrumental birth, corresponding to the rate of forceps or vacuum extractor for vaginal delivery
Oxytocin use | 10 hours
  Frequency of Oxytocin use rate after randomization.
Use of Pharmacological Analgesia for childbirth | 10 hour
  Rate of childbirth pharmacological analgesia use (including various substances and techniques such as epidural and spinal block)
Maternal fatigue level | 10 hours
  Maternal fatigue level will be evaluated using a validated questionnaire known as MATERNAL PERCEPTION OF CHILDBIRTH FATIGUE QUESTIONNAIRE (MCFQ).
  It consists of 17 items whose intensities are verified by means of a five-point score (1 to 5), with a total ranging from 17 to 85 points, in which the highest values indicate a higher level of maternal fatigue.
Maternal anxiety level | 10 hours
  Maternal anxiety during labor will be assessed using the State-Trait Anxiety Inventory (STAI).
  It consists of 19 items whose intensities are verified by means of a four-point score (1 to 4), with a total ranging from 16 to 76 points, in which the highest values indicate a higher level of anxiety.
Maternal satisfaction level | 1 hour postpartum
  The level of satisfaction with the technique (Swiss ball), reported by the participant at each assessment, may vary from zero to ten, with zero being less than satisfied and ten very satisfied with the use of the ball. Evaluated by visual analog scale (VAS).
Apgar scores | 5 minutes
  Performed in the first and fifth minutes of the child's life, the test is based on five assessment criteria: heart rate, breathing, muscle tone, reflex readiness and skin color, which, individually, can be rated from 0 to 2, totaling 10 points.
Neonatal ICU admission | 24 hour
  Rate of neonatal ICU admission according to the neonate's medical record.
Need of resuscitation of the neonate | 24 hours
  Rate of need for resuscitation of the neonate according to the neonate's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: LEILA KATZ, MD, PhD, Principal Investigator — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Delgado A, Amorim MM, Oliveira ADAP, Souza Amorim KC, Selva MW, Silva YE, Lemos A, Katz L. Active pelvic movements on a Swiss ball reduced labour duration, pain, fatigue and anxiety in parturient women: a randomised trial. J Physiother. 2024 Jan;70(1):25-32. doi: 10.1016/j.jphys.2023.11.001. Epub 2023 Nov 29. PMID 38036399